CLINICAL TRIAL: NCT03968120
Title: Effect of Lung Protective One-lung Ventilation With Fix and Variable Positive End-expiratory Pressure (PEEP) on Oxygenation and Outcome: Randomized, Controlled Trial
Brief Title: Effect of Lung Protective One-lung Ventilation With Fix and Variable PEEP on Oxygenation and Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, Head, Division General, Vascular and Thoracic Anaesthesia, University of Debrecen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DE RKEB/IKEB 4918-2017
Record Dates: First submitted 2019-05-14; First posted 2019-05-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Hypoxemia; Pulmonary Sepsis; ARDS, Human; Pneumonia
MeSH Terms: conditions — Hypoxia; Respiratory Distress Syndrome; Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Fix:One-lung ventilation with constant PEEP (No Intervention): Controll group: lung protective one-lung ventilation with fix positive end-expiratory pressure (PEEP)
- Group Variable:One-lung ventilation with variable PEEP (Active Comparator): Variable group: lung protective one-lung ventilation with variable positive end-expiratory pressure (PEEP)
  Interventions: Other: Change of ventilatory settings

INTERVENTIONS:
Other: Change of ventilatory settings — Change of Positive End-Exspiratory Pressure during one-lung ventilation
  Arms: Group Variable:One-lung ventilation with variable PEEP

SUMMARY:
During One-lung ventilation, the use of lower tidal volumes (VT) is helpful to avoid over-distension, provide sufficient oxygenation, but can result in increased atelectasis.

Nevertheless, it is not known if, during one-lung ventilation with constant low VT, moderate levels of PEEP combined with lung recruitment maneuvers are superior to variable PEEP for intraoperative oxygenation and protection against PPCs.

Aim of the study is to compare a strategy using constant tidal volume with recruitment maneuvers versus variable PEEP with recruitment maneuvers during thoracic surgery in adults.

The investigators hypothesize that in adult, non-obese patients undergoing thoracic surgery under standardized OLV with variable PEEP and recruitment maneuvers as compared to constant PEEP without recruitment maneuvers prevent PPCs.

Patients will be randomly assigned to one of two groups:

FIX PEEP VOLUME GROUP (Groupfix): mechanical ventilation with constant (6 ml/kgIBW) tidal volume and PEEP of 5 cmH2O with recruitment maneuvers

VARIABLE PEEP GROUP (Groupvar): mechanical ventilation with constant (6 ml/kgIBW) tidal volume with variable PEEP with recruitment maneuvers.

DETAILED DESCRIPTION:
Lung separation will be performed by DLT technique. Mechanical ventilation will be applied in volume-controlled mode. During two-lung ventilation, VT will be set at 8 mL/kg predicted body weight. During one-lung ventilation, in GroupFix VT will be decreased to 6 mL/kg PBW with 5 cmH2O PEEP.

In GroupVar VT mechanical ventilation with constant (6 ml/kgIBW) tidal volume with variable PEEP with recruitment maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for open thoracic or video-assisted thoracoscopic surgery under general anesthesia requiring OLV (no emergency surgery)
* BMI < 35 kg/m2
* Age ≥ 18 years
* Expected duration of surgery > 60 min
* Expected duration of anesthesia > 90 min

Exclusion Criteria:

* COPD GOLD 3+4, lung fibrosis, documented bullae, severe emphysema, pneumothorax
* uncontrolled asthma
* NYHA 3+4, CCS 3+4
* previous thoracic surgery
* ARDS (Berlin definition)
* documented pulmonary arterial hypertension > 40 mmHg syst
* documented or suspected neuromuscular disease (thymoma, myasthenia)
* planned mechanical ventilation after surgery
* bilateral procedures
* lung separation with other method than DLT (eg diff. airway, trachestomy)
* surgery in prone position
* persistent hemodynamic instability, intractable shock
* intracranial injury or tumor
* enrollment in other interventional study or refusal of informed consent
* pregnancy (excluded by anamnesis and/or laboratory analysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative oxygenation | 1 day
  PaO2 < 60 mmHg

SECONDARY OUTCOMES:
Postoperative pulmonary complications | 90 days
  Infiltrate or atelectasis on chest X-ray, fever, laboratory and physical signs of infection
Postoperative extra-pulmonary complications | 90 days
  new atrial fibrillation, tachycardia, heart failure, myocardial infarct
30 day survival/mortality | 30 days
  number of death within 30 days after surgery
90 day survival/mortality | 90 days
  number of death within 90 days after surgery
Postoperative oxygenation | 90 days
  SpO2/FiO2 ratio

CONTACTS AND LOCATIONS:
Locations (1):
- University of Debrecen, Department of Anaesthesiology and Intensive Care, Debrecen, Hungary